CLINICAL TRIAL: NCT06528639
Title: Primary Prevention Study of Cardiovascular Diseases and Diabetes in the Population With Metabolic Syndrome-A Clinical Study on Physical Exercise Guided by Cardiopulmonary Exercise Testing to Reduce the Risk of Metabolic Cardiovascular Diseases
Brief Title: A Clinical Study on Exercise Guided by CPET to Reduce the Risk of Metabolic Cardiovascular Diseases（C-MET Trial）
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: Beijing Chao Yang Hospital (Other); Guangdong Provincial People's Hospital (Other); Peking University Shenzhen Hospital (Other); The First Affiliated Hospital of Shanxi Medical University (Other); Qingdao Municipal Hospital (Other)
Responsible Party: Principal Investigator, Tang Yida, Professor, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: M2024315
Record Dates: First submitted 2024-06-27; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome; insufficient exercise
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized HIIT Group (Experimental): Participants in this group will receive a type of exercise prescription of High-Intensity Interval Training (HIIT). They will undergo supervised individualized intermittent high-intensity training (HIIT) guided by CPET three times per week under the supervision of the hospital. Participants will also receive guidance on healthy dietary habits. At the end of the 12th week, CPET and inspiratory muscle strength tests will be conducted to evaluate the training effects and adjust the exercise prescription. The total duration of the training will be 24 weeks
  Interventions: Behavioral: HIIT
- Control Group (No Intervention): Participants in this group will receive guidance on healthy dietary habits and exercise methods. They will be informed that after 24 weeks of selection, they will have the option to choose HIIT exercise program or home training.

INTERVENTIONS:
Behavioral: HIIT — Three times a week, 10 sets each session, for 24 weeks of high-intensity interval training.
  Arms: Individualized HIIT Group

SUMMARY:
The main purpose of this study is to validate the effect of an individualized exercise prescription developed based on cardiopulmonary exercise testing (CPET) in subjects with metabolic syndrome. This study aims to assess the improvement in cardiovascular metabolic risk associated with the personalized exercise regimen,known as individualized HIIT.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 30 and 65, for both males and females;
2. Inadequate exercise: Sedentary lifestyle: Sitting for more than 6 hours daily over the past 6 months; Insufficient physical activity evaluated by the International Physical Activity Questionnaire (IPAQ), with an average weekly duration of moderate-intensity physical activity less than 150 minutes or high-intensity physical activity less than 75 minutes;
3. Meeting the criteria for metabolic syndrome according to the 2009 AHA/IDF definition: Must have three or more of the following: Abdominal obesity(Waist circumference ≥90 cm for males, ≥80 cm for females); Elevated fasting blood glucose: ≥5.6 mmol/L; Elevated blood pressure: Systolic blood pressure ≥130 mm Hg, or diastolic blood pressure ≥85 mm Hg; Elevated fasting triglycerides (TG): ≥1.7 mmol/L (150 mg/dl); Reduced fasting high-density lipoprotein cholesterol (HDL-C): <1.0 mmol/L for males, <1.3 mmol/L for females.

   Additionally, must meet the following conditions: TG <500 mg/dl (5.6 mmol/L); fasting blood glucose <7 mmol/L; baseline blood pressure <140/90 mm Hg;
4. Willingness to improve health status through reasonable exercise.

Exclusion Criteria:

1. Contraindications to CPET (Cardiopulmonary Exercise Testing);
2. Positive results in CPET exercise electrocardiogram;
3. The patient has elevated LDL-C levels and has been indicated for statin therapy.
4. Currently undergoing treatment with antihypertensive, antidiabetic, lipid-lowering, or antiarrhythmic medications;
5. The doctor evaluates dietary supplements or over-the-counter medications that may affect the results (such as fish oil products, red yeast rice extract, over-the-counter weight loss drugs, meal replacements, probiotics, berberine, etc.)
6. Mental disorders;
7. Conditions related to exercise impairment, or occurrence of lower limb exercise-related injuries in the past 6 months;
8. Women who are pregnant, breastfeeding, or planning to become pregnant in the near future;
9. Other situations deemed unsuitable for participation in this study by the researchers;
10. Refusal to sign the informed consent form.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in composite cardiovascular disease risk score (z-score) | through study completion, an average of 2 year
  The primary outcome is the change from baseline in the composite cardiovascular disease risk score (z-score) calculated using resting blood pressure, high-density lipoprotein cholesterol, fasting glucose, waist circumference and triglyceride. Each risk factor will be individually standardized and expressed as sex-specific z-score by using the formula = (value - mean)/standard deviation for each participant.

SECONDARY OUTCOMES:
Biochemical and metabolic indicators | through study completion, an average of 2 year
  Biochemical indicators including GLU(mmol/L),CHO(mmol/L),TG(mmol/L),LDL-C(mmol/L),HDL-C(mmol/L) etc.
CPET (Cardiopulmonary Exercise Testing) related indicators | through study completion, an average of 2 year
  Peak oxygen uptake（ml/min）
calf circumference, waist circumference, and hip circumference | through study completion, an average of 2 year
  Indicators in terms of length include: calf circumference, waist circumference, and hip circumference
Oral Glucose Tolerance Test (OGTT) Related Indicators | through study completion, an average of 2 year
  Fasting Blood Glucose and Insulin, 30-minute Postprandial Blood Glucose and Insulin, 120-minute Postprandial Blood Glucose and Insulin.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Da Tang, MD, PhD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No